CLINICAL TRIAL: NCT03775876
Title: Dexmedetomidine Versus Propofol in Conjunction With Regional Block for Shoulder Arthroscopy: a Randomized Controlled Double Blind Trial
Brief Title: Dexmedetomidine Versus Propofol in Conjunction With Regional Block for Shoulder Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Hicham Abou Zeid, Assistant Professor, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CEHDF 945
Record Dates: First submitted 2018-11-18; First posted 2018-12-14 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Hemodynamic; Sedation; Satisfaction, Personal
Keywords: Propofol; Dexmedetomidine; Regional anesthesia; Satisfaction; Shoulder arthroscopy
MeSH Terms: conditions — Personal Satisfaction | interventions — Surgical Procedures, Operative; Propofol; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: randomised controlled double blind trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: surgeons, patients as well as the outcome assessor were blinded in regards of the drug used for sedation during surgery (Propofol vs dexmedetomidine)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Patients programmed for elective Shoulder arthroscopy surgery will receive a continuous intravenous infusion of Propofol. Infusion will be started after regional block (interscalene) being performed and will be continued to the end of wound closure. Infusion will be started at 2mg/Kg/h and modified to a maximum of 4 mg/Kg/h in order to achieve a bispectral index (BIS) between 60 and 90 and a Ramsay sedation score between two and four.
  Interventions: Procedure: Shoulder Arthroscopy; Procedure: Regional Block; Drug: Propofol; Diagnostic Test: BIS
- Dexmedetomidine (Active Comparator): Patients programmed for elective Shoulder arthroscopy surgery will receive a continuous intravenous infusion of Dexmedetomidine. Infusion will be started after regional block (interscalene) being performed and will be continued to the end of wound closure. Infusion will be started at 1mcg/kg over 10 minutes then 0.2 mcg/Kg/h and modified to a maximum of 0.7 mcg/Kg/h in order to achieve a bispectral index (BIS) between 60 and 90 and a Ramsay sedation score between two and four with a maximum.
  Interventions: Procedure: Shoulder Arthroscopy; Procedure: Regional Block; Drug: Dexmedetomidine; Diagnostic Test: BIS

INTERVENTIONS:
Procedure: Shoulder Arthroscopy — patients in both groups are programmed for an elective shoulder arthroscopy surgery
  Other Names: Surgery
Procedure: Regional Block — patients in both groups received regional block for anesthesia: brachial plexus blockade was performed using the interscalene approach under ultrasound combined to nerve stimulation. 20 ml ropivacaine 0.375% were injected.
  Other Names: Interscalene brachial plexus block
Drug: Propofol — propofol 10mg/ml was used for sedation as described in the arms section
  Other Names: Propofol-Lipuro
  Arms: Propofol
Drug: Dexmedetomidine — Dexmedetomidine was diluted to 4mcg/ml and used for sedation as described in the arms section
  Other Names: Dexmedetomidine Hcl 100 mcg (Micrograms)/ml Inj
  Arms: Dexmedetomidine
Diagnostic Test: BIS — sedation level was monitored using bispectral index to achieve values described in the arms group
  Other Names: Bispectral index

SUMMARY:
Operative shoulder arthroscopy under regional block anesthesia often presents with hemodynamic challenges for the anesthesiologist, knowing that a low systolic blood pressure is required to minimize the bleeding. Regional anesthesia is successfully performed to many patients in whom tracheal intubation or the placement of a laryngeal tube is undesired. Propofol has traditionally been used to provide sedation in patients undergoing shoulder arthroscopy under regional anesthesia. In contrast to Propofol, Dexmedetomidine is a highly selective α-2 adrenoceptor agonist that has been shown to provide sedation, analgesia and anxiolytic effects with minimal respiratory depression. Due to the effect of both drugs on blood pressure, the investigators set out to compare intraoperative hemodynamics of both drugs, along with the surgeon's satisfaction and the degree of comfort provided to patients undergoing interscalene brachial plexus block for shoulder arthroscopy. The investigators also assessed whether the type of anesthetic agent used for sedation accounted for other differences in intra and post-operative outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists score (ASA) I or II.
* Elective Shoulder arthroscopy.

Exclusion Criteria:

* Allergies to any of the used medications.
* ASA score of III or above.
* Cardiac abnormalities.
* Contraindications to regional blocks.
* Patient refusal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
iSBP | Hour 0
  initial Systolic Blood Pressure (iSBP) measurement at arrival to the operating room. Hour 0 is the time of patient's arrival to the operating room.
iMAP | Hour 0
  initial Mean Arterial blood Pressure (iMAP) measurement at arrival to the operating room. Hour 0 is the time of patient's arrival to the operating room.
SBP | at 10 minutes interval from the beginning up to 0 minutes after the end of Propofol or Dexmedetomidine infusion
  Change in Systolic Blood Pressure from iSBP
MAP | at 10 minutes interval from the beginning up to 0 minutes after the end of Propofol or Dexmedetomidine infusion
  change in Mean Arterial blood Pressure from iMAP
Surgeon Satisfaction: Global satisfaction scale | up to 1 hour after surgery completion
  Global satisfaction of the surgeon regarding anesthesia and patient immobility on a scale from 0 (not satisfied) to 10 (completely satisfied) collected at the end of surgery
Estimation of Bleeding | up to 1 hour after surgery completion
  Surgeon's evaluation of the bleeding that had affected the surgeon's visibility on a scale from 0 (no bleeding) to 5 (very intense bleeding) collected at the end of surgery
Occurence of Hypotension | up to 0 minutes after admission to the Post Anesthesia Care Unit (PACU)
  number of episodes of hypotension ( a drop of systolic blood pressure >30% of the initial value recorded at patient arrival to the operating theatre)

SECONDARY OUTCOMES:
RR | at 10 minutes interval from the beginning up to 0 minutes after the end of Propofol or Dexmedetomidine infusion
  respiratory rate (RR) per minute
BPM | at 10 minutes interval from the beginning up to 0 minutes after the end of Propofol or Dexmedetomidine infusion
  Beats per minute (BPM)
SaO2 | at 10 minutes interval from the beginning up to 0 minutes after the end of Propofol or Dexmedetomidine infusion
  Oxygen Saturation (SaO2) (%)
Vasopressors OR | up to 0 minutes after admission to the PACU
  use of vasoactive drugs during surgery (Yes or No)
Vasopressors PACU | up to 3 hours after surgery completion
  use of vasoactive drugs during PACU stay (Yes or No)
tBIS | up to 0 minutes after the end of Propofol or Dexmedetomidine infusion
  time to achieve desired Bispectral Index (tBIS) level (minutes)
PS1: scale | up to 3 hours after surgery completion
  Patient Satisfaction 1(PS1): I would want to have the same anesthetic again on a 5 points Likert scale from 0 to 4: 0= Strongly disagree, 1= Disagree, 2= Neither agree nor disagree, 3= Agree, 4= Strongly agree.
PS2: scale | up to 3 hours after surgery completion
  Patient Satisfaction 2(PS2): I felt pain on a 5 points Likert scale from 0 to 4: 0= Strongly disagree, 1= Disagree, 2= Neither agree nor disagree, 3= Agree, 4= Strongly agree.
PS3: scale | up to 3 hours after surgery completion
  Patient Satisfaction 3(PS3): I was satisfied with my anesthetic care on a 5 points Likert scale from 0 to 4: 0= Strongly disagree, 1= Disagree, 2= Neither agree nor disagree, 3= Agree, 4= Strongly agree.
PS4: scale | up to 3 hours after surgery completion
  Patient Satisfaction 4(PS4): I felt relaxed during the procedure on a 5 points Likert scale from 0 to 4: 0= Strongly disagree, 1= Disagree, 2= Neither agree nor disagree, 3= Agree, 4= Strongly agree.
PON | up to 3 hours after surgery completion
  Occurrence of Post Operative Nausea (PON) at PACU at least on episode (yes or No)
POV | up to 3 hours after surgery completion
  Occurence of Post Operative Vomiting (POV) at PACU at least on episode (yes or No)
Need for rescue analgesia: RA | up to 3 hours after surgery completion
  need for rescue analgesia (RA) opioids at PACU (Yes or No)
ALDRETE score | up to 3 hours after surgery completion
  time to reach modified Aldrete score of 9/10 at PACU (minutes)
VASi | up to 10 minutes after admission to the PACU
  Visual Analog Scale initial (VASi): Visual analog rating scale for pain (VAS) in which 0 is defined as no pain and 10 as maximum pain at PACU arrival (0-10)
VASd | up to 3 hours after surgery completion
  Visual Analog Scale discharge (VASd): Visual analog rating scale for pain in which 0 is defined as no pain and 10 as maximum pain at PACU discharge (0-10)
Occurence of Bradycardia | up to 0 minutes after admission to the PACU
  number of episodes of bradycardia (Heart rate <45/min)

OTHER OUTCOMES:
BIS level | at 10 minutes interval from the beginning up to 0 minutes after the end of Propofol or Dexmedetomidine infusion
  Bispectral index (BIS) level value (0-100). BIS is used to monitor depth of anesthesia or sedation.The BIS is an electroencephalogram-derived multivariant scale.The BIS monitor provides a single dimensionless number, which ranges from 0 (equivalent to EEG silence) to 100 (Normal EEG activity or patient completely awake). 0 = EEG silence, [0 to 20] = burst suppression on EEG, [20 to 40] = deep hypnotic state, [40 to 60] = general anesthesia, [60 to 80] = sedation but individual responds to loud commands or mild shaking, [80 to 99] = sedation but individual responds to normal voice and 100 = Completely Awake.
Ramsay sedation scale | at 10 minutes interval from the beginning up to 0 minutes after the end of Propofol or Dexmedetomidine infusion
  Ramsay sedation scale value (1-6): 1=Anxious, agitated, restless; 2=Cooperative, oriented, tranquil; 3=Responsive to commands only; 4=Brisk response to light glabellar tap or loud auditory stimulus; 5=Sluggish response to light glabellar tap or loud auditory stimulus; 6=No response to light glabellar tap or loud auditory stimulus.
Sedation Duration | up to 0 minutes after the end of Propofol or Dexmedetomidine infusion
  total duration of Propofol or Dexmedetomidine infusion in minutes
Sedation Dose | up to 0 minutes after the end of Propofol or Dexmedetomidine infusion
  total dose of Propofol (mg) or Dexmedetomidine (mcg) used

CONTACTS AND LOCATIONS:
Overall Officials: Hicham A ABOU ZEID, M.D., M.Sc., Study Chair — Saint Joseph University School of Medicine; Nouhad S AYOUB, M.D., Principal Investigator — Saint Joseph University School of Medicine
Locations (1):
- Hotel Dieu de France Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peng K, Li J, Ji FH, Li Z. Dexmedetomidine compared with propofol for pediatric sedation during cerebral angiography. J Res Med Sci. 2014 Jun;19(6):549-54. PMID 25197298
- [Background] Kim N, Yoo YC, Lee SK, Kim H, Ju HM, Min KT. Comparison of the efficacy and safety of sedation between dexmedetomidine-remifentanil and propofol-remifentanil during endoscopic submucosal dissection. World J Gastroenterol. 2015 Mar 28;21(12):3671-8. doi: 10.3748/wjg.v21.i12.3671. PMID 25834336
- [Background] Wu Y, Zhang Y, Hu X, Qian C, Zhou Y, Xie J. A comparison of propofol vs. dexmedetomidine for sedation, haemodynamic control and satisfaction, during esophagogastroduodenoscopy under conscious sedation. J Clin Pharm Ther. 2015 Aug;40(4):419-25. doi: 10.1111/jcpt.12282. Epub 2015 May 13. PMID 25970229